CLINICAL TRIAL: NCT05142566
Title: Prospective Multicenter MANTA™ Vascular Closure Device Ultrasound Guided Closure Study
Brief Title: MANTA Ultrasound Closure Study
Acronym: MANTA ULTRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Ineffective enrollment
Sponsor: Essential Medical, Inc. (Industry)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-3370
Record Dates: First submitted 2021-11-10; First posted 2021-12-02 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: Femoral Arteriotomy Closure
Keywords: MANTA; Arterial Closure Device; Ultrasound Closure; Large Bore Closure Device

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ultrasound Closure (Experimental): Open label, single arm study using ultrasound guidance during MANTA device deployment.
  Interventions: Device: MANTA Vascular Closure Device

INTERVENTIONS:
Device: MANTA Vascular Closure Device — Evaluate the safety of ultrasound guided deployment of MANTA VCD.

SUMMARY:
Demonstrate the safety of MANTA Vascular Closure Device (VCD) ultrasound (U/S) guided closure in patients undergoing elective TAVR procedures with planned percutaneous femoral arterial access.

DETAILED DESCRIPTION:
The MANTA Vascular Closure Device is indicated for closure of femoral arterial access sites while reducing time to hemostasis following the use of 10-20F devices or sheaths (12-25F OD) in endovascular catheterization procedures.

This study is being conducted to demonstrate the safety of U/S guided closure with MANTA VCD following TAVR procedures utilizing large bore sheaths.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for elective or planned (i.e., not emergent or urgent) percutaneous transcatheter valve replacement (TAVR) via a 10-20F device or sheath (12-25F OD) with common femoral artery approach
* Vessel size would allow for access for the MANTA VCD based on vessel size as determined by baseline CTA: minimum vessel diameter of 5mm for the 14F MANTA VCD and 6mm for the 18F MANTA VCD
* Understand and sign the study specific written informed consent form and PHI authorization
* Able and willing to fulfill the follow-up requirements

Exclusion Criteria:

* Patients known to be pregnant or lactating
* Patients who have a systemic infection or a local infection at or near the access site
* Patients with significant anemia (hemoglobin ≤10 g/DL)
* Patients who are morbidly obese or cachectic (BMI >40 or <20kg/m2)
* Patients with a known bleeding disorder including thrombocytopenia (platelet count <100,000 cells/UL), thrombasthenia, hemophilia, or von Willebrand disease
* Patients with allergy to bovine materials or any other device material, including collagen and/or collagen products, polyglycolic or polylactic acid, stainless steel or nickel
* Patients with a femoral artery puncture in target groin within the prior 30 days, prior vascular closure device placement in the target common femoral artery within 3 months, or any prior target femoral artery access-related complication
* Patients who have undergone use of an intra-aortic balloon pump (IABP) through the arterial access site within 30 days prior to the baseline evaluation.
* Patients who have a Common Femoral Artery (CFA) with visible calcium and/or tortuosity, as determined by baseline CTA, precluding safe access and likely to interact with large bore access site arteriotomy, determined by investigator.
* Patients with previous iliofemoral intervention in region of access site, including but not limited to prior atherectomy, stenting, surgical or grafting procedures in the access area
* Patients in whom oral anticoagulation therapy cannot be stopped for the peri procedural period or patients with INR >1.8 at the time of the procedure
* Patients who are unable to ambulate at least 6 meters without assistance at baseline
* Patients with renal insufficiency (serum creatinine >2.5 mg/dl) or on dialysis therapy
* Patients with existing nerve damage in the ipsilateral leg
* Patients with a further planned endovascular procedure within the next 30 days
* Patients who have already participated in this IDE study
* Patients who are currently participating in another clinical study of an unapproved investigational device or drug that has not concluded the follow-up period or patient currently participating in another clinical study likely to influence hemostasis and vascular complications
* Patients who cannot adhere to or complete the investigational protocol for any reason including but not limited to geographical residence, psychiatric condition or life threatening disease
* Patients who have a common femoral artery <5mm in diameter for the 14F MANTA VCD or <6 mm in diameter for the 18F MANTA VCD, common femoral artery stenosis resulting in a vessel diameter <5mm in diameter for the 14F MANTA VCD or <6 mm in diameter for the 18F MANTA VCD, or > 50% diameter femoral or iliac artery stenosis
* Patients in whom, during initial access of the artery, arteriotomy and surrounding anatomy cannot be visualized and identified clearly under U/S imaging and/or if the vertical depth from the surface of the skin to target area of the common femoral artery measures greater than 6cm

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wood, Principal Investigator — Vancouver General Hospital; Vijay Iyer, Principal Investigator — University at Buffalo
Locations (6):
- United States (5):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Henry Ford, Detroit, Michigan
  - University of Buffalo, Buffalo, New York
  - Baylor Scott & White, Round Rock, Texas
  - Sentara Northern Virginia Medical Center, Woodbridge, Virginia
- Vancouver General Health, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data obtained will be used, without mentioning Subject PHI, to assess the results of the research, and the data could be used in the future with regard to this study or other studies. The data can be passed on to the health authorities for the purposes of registering the medical device.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: one subject was treated by a physician who was not officially trained and signed off on the protocol or device.
Period: Overall Study
Arm/Group | Ultrasound Closure
Started | 18
Completed | 17
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 80.06 [69 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 11
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Any Large Bore Access-site Related VARC-2 Major Vascular Complication
Description: adapted from VARC-2 Criteria
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Participants | 0

2. Secondary Outcome: Time to Hemostasis
Description: The elapsed time between VCD deployment and first observed and confirmed arterial hemostasis.
Time Frame: During the procedure
Measure: Median (Full Range); unit: Minutes
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Minutes | .42 [0.00 to 9.87]

3. Secondary Outcome: Number of Patients With Technical Success
Description: Percutaneous vascular closure is obtained without the use of unplanned endovascular or surgical intervention.
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Participants | 17

4. Secondary Outcome: Number of Subjects With Ambulation Success
Description: If a previously ambulatory patient (until day of TAVI) is able to ambulate for at least 20 feet/6 meters without re-bleeding.
Time Frame: During procedure admission
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Participants | 17

5. Secondary Outcome: Time to Ambulation
Description: The elapsed time between VCD deployment and when ambulation is achieved.
Time Frame: During procedure admission
Measure: Median (Full Range); unit: hours
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
hours | 8.93 [4.21 to 119.05]

6. Secondary Outcome: Treatment Success
Description: Time to Hemostasis ≤10 minutes and no VACR-2 Major complications
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Participants | 17

7. Secondary Outcome: Procedure Time
Description: Elapsed time from initial skin break to time when the post-deployment angiogram is completed.
Time Frame: During the procedure
Measure: Median (Full Range); unit: Hours
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Hours | 0.75 [0.61 to 1.62]

8. Secondary Outcome: Rate of Any Large Bore Access-site Related VARC-2 Minor Vascular Complication
Description: adapted from VARC-2 Criteria
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound Closure
Number analyzed (Participants) | 17
Participants | 1

ADVERSE EVENTS:
Time Frame: Index procedure up to 30 days
Arm/Group | Ultrasound Closure
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Closure (N=17)
Transient Ischemic Attack (TIA) (Nervous system disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Systemic Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Closure (N=17)
Access Site Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Vessel Dissection (Vascular disorders) | 1 (1)
Edema in left hand (Vascular disorders) | 1 (1)
Retroperitoneal Bleed (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The Prospective Multicenter MANTA™ Vascular Closure Device Ultrasound Guided Closure Study (ST-3370) was terminated early primarily for business reasons. The sponsor recognized that the conditions for widespread adoption of ultrasound-based MANTA deployment do not presently exist. As a result of this finding and the likelihood that the study would not provide sufficient data to support a future labeling change, the sponsor decided to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT05142566/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT05142566/SAP_001.pdf